CLINICAL TRIAL: NCT06548139
Title: Multicenter, Randomized, Double-blind, Positive Control Evaluation of Rabies Monomab CBB 1 Combination Vaccine for Antibody Neutralization Activity and Safety Phase Clinical Trials in Healthy People
Brief Title: Rabies mAb CBB 1 Combination Vaccine in Healthy People With Antibody Neutralization Activity and Safety Phase Clinical Trials
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changchun BCHT Biotechnology Co. (Industry)
Collaborators: The First Affiliated Hospital of Yunnan University of Traditional Chinese Medicine (Unknown); Anning City First People's Hospital (Unknown); Yunnan Central Hospital (Unknown); Beijing Contreke Statistical Technology Co., LTD (Unknown); Military Science Zhengyuan (Beijing) Pharmaceutical Research Co., LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B1801-F20220212
Record Dates: First submitted 2024-07-16; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-07

CONDITIONS: Rabies Virus Infection
Keywords: Rabies Virus Neutralizing Antibodies; Safety; Immunogenicity
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Intervention Model Description: There were 120 healthy people aged 10-50 years, divided into 3 groups: test group 1 rabies mAb CBB1 50.0 µ g / kg + vaccine; test group 2 rabies mAb CBB1 100.0 µ g / kg + vaccine; and control group HRIG 20IU / kg + vaccine
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): Natural full human monoclonal antibody CBB 1 injection：Each dose (2.5ml) contained 0.5 mg / natural monoclonal antibody ml CBB 1 Ingredients: 25 mM citrate buffer, 125 mM sodium chloride, 0.02% (w / v) polysorbate 20 and water for injection Character: colorless to pale green and yellow liquid Specification: 1.25 mg (2.5 ml) / bottle Mode of administration: intramuscular injection of the vastus lateralis muscle. Usage and dosage: The injection dose was calculated according to the group and body weight of the volunteer. On day 0, unilateral or bilateral extrafemoral muscle group injections were selected by dose, with no more than 5 mL at each site, and at least 2.5 cm apart.
  Interventions: Drug: Natural full human monoclonal antibody CBB 1 injection 50.0µg/kg; Biological: Lyophilized rabies vaccine for human use (Vero cells)
- Experimental group 2 (Experimental): Natural full human monoclonal antibody CBB 1 injection：Each dose (2.5ml) contained 0.5 mg / natural monoclonal antibody ml CBB 1 Ingredients: 25 mM citrate buffer, 125 mM sodium chloride, 0.02% (w / v) polysorbate 20 and water for injection Character: colorless to pale green and yellow liquid Specification: 1.25 mg (2.5 ml) / bottle Mode of administration: intramuscular injection of the vastus lateralis muscle. Usage and dosage: The injection dose was calculated according to the group and body weight of the volunteer. On day 0, unilateral or bilateral extrafemoral muscle group injections were selected by dose, with no more than 5 mL at each site, and at least 2.5 cm apart.
  Interventions: Drug: Natural full human monoclonal antibody CBB 1 injection 100.0µg/kg; Biological: Lyophilized rabies vaccine for human use (Vero cells)
- Positive control group (Active Comparator): Rabies Human Immunoglobulin (HRIG) Active ingredient: Rabid human immunoglobulin Specification: 200 IU / 2 ml / bottle Administration mode: intramuscular injection of the vastus lateral muscle group.
  Usage and dosage: the injection dose was calculated according to the body weight of the volunteer. On day 0, unilateral or bilateral extrafemoral muscle group injections were selected by dose, with no more than 5 mL at each site and at least 2.5 cm apart
  Interventions: Drug: Rabies Human Immunoglobulin (HRIG); Biological: Lyophilized rabies vaccine for human use (Vero cells)

INTERVENTIONS:
Drug: Natural full human monoclonal antibody CBB 1 injection 50.0µg/kg — Active ingredient: natural full human monoclonal antibody CBB 1 containing 0.5 mg / ml per dose (2.5ml) Ingredients: 25 mM citrate buffer, 125 mM sodium chloride, 0.02% (w / v) polysorbate 20 and water for injection
  Arms: Experimental group 1
Drug: Natural full human monoclonal antibody CBB 1 injection 100.0µg/kg — Active ingredient: natural full human monoclonal antibody CBB 1 containing 0.5 mg / ml per dose (2.5ml) Ingredients: 25 mM citrate buffer, 125 mM sodium chloride, 0.02% (w / v) polysorbate 20 and water for injection
  Arms: Experimental group 2
Drug: Rabies Human Immunoglobulin (HRIG) — Active ingredient: Rabid human immunoglobulin
  Arms: Positive control group
Biological: Lyophilized rabies vaccine for human use (Vero cells) — Active ingredient: inactivated rabies virus fixed poison

SUMMARY:
To evaluate the antibody neutralization activity and safety of rabies mAb CBB 1 combination vaccine used in healthy people

DETAILED DESCRIPTION:
To evaluate the rabies virus neutralizing antibody (RVNA) activity of rabies mAb CBB 1 in combination with human rabies vaccine (Vero cells) in healthy volunteers.

To evaluate the safety and tolerability of rabies mAb CBB 1 compared to HRIG in combination with human rabies vaccine (Vero cells) in healthy volunteers.

To evaluate the immunogenicity of rabies mAb CBB 1.

ELIGIBILITY:
Inclusion Criteria:

1. Before the trial, I have had a detailed understanding of the nature, significance and possible benefits of the trial, the possible inconvenience and potential risks and discomfort, and volunteered to participate in this clinical trial, was able to communicate well with researchers, comply with the requirements of the whole study, and signed a written informed consent;
2. Men or women aged 18~50 (including boundary values) at the time of screening;
3. The weight of female volunteers was 45.0 kg and 80.0 kg, that of male volunteers was 50.0 kg and 80.0 kg, and the body mass index (BMI) was between 18.0 and 27.0 kg/m2 (including boundary value) (BMI= weight kg / height m2);
4. Female volunteers have no fertility or egg donation plan within 14 days before the first dose to 3 months after the end of the trial and voluntarily take effective physical contraception, while male volunteers have no fertility or sperm donation plan within 3 months after the first dose to the trial and voluntarily take effective physical contraception.

Exclusion Criteria:

1. Those who are known to be allergic to the study drug (including excipients, similar drugs), or suffer from severe allergic diseases or allergic constitution (such as allergic to two or more drugs, food or pollen), may damage the safety of the volunteers in the judgment of the investigator (inquiry);
2. Those with a clear history of allergy to the essential substances (such as skin disinfectants) that may be exposed to during the test (inquiry);
3. Patients with a history of clinically serious disease within 6 months (180 days) before the first dose and not cured, or patients with acute or chronic diseases that may significantly affect the in vivo process or safety evaluation of the study drug (inquiry);
4. Patients with a previous history of autoimmune diseases or chronic hepatitis (inquiry);
5. Patients with a previous history of convulsions, epilepsy, mental or nervous system, or a family history of convulsions or epilepsy (inquiry);
6. Those who have received major surgery within 3 months (90 days) prior to the first dose, or those who may significantly affect the internal process or safety evaluation of the study drug (inquiry, inquiry);
7. Patients with a history of rabies virus infection or have received rabies vaccination (inquiry);
8. Suspected or clear identification of a history of injuries to warm-blooded mammals in the last 12 months (360 days) (warm-blooded animals refer to animals that can regulate their body temperature, also known as endotherms. Birds and the vast majority of mammals, including the cats and dogs around them, are warm-blooded animals) (inquiry);
9. Having received a vaccine other than the rabies vaccine within 1 month (30 days) prior to the first dose (inquiry);
10. Those who have used a rabies passive immunization preparation or used systemic immunosuppressive agents such as glucocorticoids within 3 months (90 days) prior to the first dose (inquiry, inquiry)；
11. Those who have been used or are in the current period) or who may have a significant impact on the in vivo process or safety evaluation of the study drug (inquiry, inquiry);
12. Any clinical trial drug or device used within 3 months (90 days) prior to the first dose, or <5 half-lives of the last previous trial drug dose (whichever is older), or planned to participate in other clinical trials during the study (inquiry, inquiry);
13. Regular alcohol for 3 months (90 days) before the first dose (3 times a week, and an average of 50° of liquor 200 ml) (inquiry);
14. Those with positive alcohol breath test or test value> 0 mg / 100 ml (examination);
15. Cigarette addiction (more than 10 cigarettes or the same amount of tobacco per day) within 1 month (30 days) before the first dose (inquiry);
16. Those who lost blood / donated more than 400 ml (other than female physiological blood loss) within 3 months (90 days) before the first dose, or who received blood transfusion or used blood products, or planned to donate blood during the trial or within 1 month (30 days) after the end of the trial (inquiry);
17. Those who ingested alcohol-containing products within 24 hours before the first dose (inquiry);
18. Abnormalities at the administration site (such as inflammation, induration, redness, large area scar or tattoo, etc.) shall affect the administration or the clinical observer (examination);
19. Those with a history of substance abuse (inquiry);
20. Those who are screened positive for substance abuse during the screening period (examination);
21. Those who are positive for the initial HIV screening during the screening period (screening);
22. two half and half qualitative tests of hepatitis B during the screening period (examination);
23. Patients with positive results for hepatitis C virus antibody or treponema pallidum antibody during the screening period (examination);
24. Physical examination, vital signs (respiration, blood pressure, pulse rate), electrocardiogram, other laboratory tests (laboratory tests not listed separately) or other auxiliary examination results are judged as abnormal and clinically significant by the study doctor (examination);
25. Ear temperature during the screening period is> 37.5℃ (examination);
26. Women who are positive in pregnancy or lactation or screening pregnancy test (inquiry, examination);
27. Patients with a history of needle acupuncture, blood sickness, or unable to tolerate venipuncture (inquiry);
28. The volunteers may be unable to cooperate with the study for other reasons or the investigators is not unsuitable for inclusion.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Rabia for neutralizing antibody activity | 7 Days
  Geometric mean RVNA concentration on day 7 after medication; Proportion of volunteers with 0.5 IU / ml of RVNA on day 7 after medication.

SECONDARY OUTCOMES:
Rabia for neutralizing antibody activity | 105 Days
  RVNA detection rate at days 0.5,1,2,3,5,7,14,28,42,84, and 105 after drug administration.
  Geometric mean concentration and relative antibody positive rate at days 0.5,1,2,3,5,105,28,42,84,105 (RVNA 0.5 IU / ml).
Safety evaluation index | 105 Days
  Clinical indicators:Physical examination.
Safety evaluation index | 105 Days
  Vital signs: ear temperature/℃
Safety evaluation index | 105 Days
  Vital signs: blood pressure (sitting position)/mmHg
Safety evaluation index | 105 Days
  Vital signs: pulse rate/Time / minute.
Safety evaluation index | 105 Days
  12-lead ECG all were abnormal and clinically significant by the investigator
Safety evaluation index | 105 Days
  local reaction;constitutional reaction.
Safety evaluation index | 105 Days
  Laboratory indicator all were abnormal and clinically significant by the investigator
Immunogenicity evaluation index | 105 Days
  Positive rate of anti-drug antibodies (ADA) on days 14,28,84,105 after administration. If ADA positive, continue to evaluate whether it is rabies mAb CBB 1 neutralizing antibody

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Yunnan University of Traditional Chinese Medicine, Kunming, Yunnan, China